CLINICAL TRIAL: NCT06308484
Title: Neuromodulation and Mindfulness as Therapeutic Treatment in Detoxified Patients With AUD
Brief Title: Neuromodulation and Mindfulness Patients With AUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Medical School Berlin (Other)
Responsible Party: Principal Investigator, Anne Beck, Prof. Dr. Anne Beck, Health and Medical University Potsdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TRR265 C02 FP2
Record Dates: First submitted 2024-02-26; First posted 2024-03-13 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active transcutaneous vagus nerve stimulation (Active Comparator): The tVNS device consisted of two titan electrodes mounted on a gel frame and connected to a wired neurostimulation device (tVNS Health GmbH, Germany). Electrodes were placed on the cymba conchae. Stimulation intensity of 0.5 mA, delivered with a pulse width of 200-300 μs at 25 Hz.
  Interventions: Device: Transcutaneous vagus nerve stimulation
- Sham transcutaneous vagus nerve stimulation (Sham Comparator): Stimulation parameters equivalent to active but sham stimulation was administered by positioning the electrodes on the central part of the left earlobe rather than the outer auditory canal, as the earlobe lacks vagus innervation.
  Interventions: Device: Transcutaneous vagus nerve stimulation
- Closed-loop AM-tACS increase frontal midline theta oscillation (Active Comparator): We will deliver amplitude-modulated transcranial alternating current stimulation (AM-tACS) using two circular rubber electrodes (4 cm diameter) positioned at the Fpz and Cz locations of the international 10-20 system. The AM-tACS stimulation waveform features a carrier signal frequency of 10 kHz, an amplitude of ±1 mA, and a signal that is real-time synchronized with theta oscillations of the frontal midline. In the active condition target oscillations (frontal midline theta) will be increased.
  Interventions: Device: Closed-loop AM-tACS
- Closed-loop AM-tACS decrease frontal midline theta oscillation (Sham Comparator): Equivalent to the active comparator - except here the target oscillation will be suppressed.
  Interventions: Device: Closed-loop AM-tACS

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation — Patients that are enrolled in a MBRP program will be subjected to weekly tVNS stimulation during a 30-minute audio guided mindfulness exercise.
  Arms: Active transcutaneous vagus nerve stimulation; Sham transcutaneous vagus nerve stimulation
Device: Closed-loop AM-tACS — Patients that are enrolled in a MBRP program will be subjected to weekly CLAM-tACS stimulation during a 30-minute audio guided mindfulness exercise.
  Arms: Closed-loop AM-tACS decrease frontal midline theta oscillation; Closed-loop AM-tACS increase frontal midline theta oscillation

SUMMARY:
Our primary objective is to integrate tVNS and mindfulness meditation within a structured mindfulness-based relapse prevention (MBRP) program for detoxified alcohol-dependent patients (AD). We aim to determine whether neuromodulation can enhance mindfulness-based relapse prevention compared to mindfulness practice alone. In this context, we will investigate potential changes in the interaction of top-down control and cue reactivity, as well as assess the severity of AUD. Measurements of drinking behavior, cravings, and abstinence rates will be conducted up to three months post-treatment. Our second objective is to examine the causal role of frontal midline theta oscillations (FMΘ) in MBRP and cognitive control. To achieve this, we will first establish closed-loop amplitude-modulated transcranial alternating current stimulation (CLAM-tACS) to selectively modulate FMΘ oscillations during MBRP meditation exercises in AUD patients (2).

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Dependence (ICD-10)
* abstinence between 3 days and 12 months

Exclusion Criteria:

* current (last 12 months) substance use disorder/dependence
* neurological disorders (e.g. epilepsy, neuropathy, multiple sclerosis)
* current severe major depressive disorder, manic episode or schizophreniform disorder
* intake of anticonvulsive or high-potency antipsychotic medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Control | Pre and post intervention after 6-8 weeks
  Before and after the treatment, we will assess cognitive control on a behavioral (response inhibition) and neurophysiological level (electroencephalogram) using a Simon GoNogo task, which reliably triggers activation of the frontal midline regions (Swick et al., 2011).
Interoception | Pre and post intervention after 6-8 weeks
  Additionally, interoceptive control is intended to be measured using a heartbeat detection task (Kleckner et al., 2015).
Cue-Reactivity | Pre and post intervention after 6-8 weeks
  Evaluate physiological reactivity to alcohol cues through a passive viewing task developed based on the guidelines of Ekhitiari et al. (2022) and measure subjective cue-induced cravings.

SECONDARY OUTCOMES:
Heartrate | pre, ad interim at every tVNS and CLAM-tACS stimulation (once per week for 6-8 weeks), post after 6-8 weeks
  Heartrate change due to stimulation
Heartrate Variability | pre, ad interim at every tVNS and CLAM-tACS stimulation (once per week for 6-8 weeks), post after 6-8 weeks
  Heartrate variability change due to stimulation
Mindfulness | pre, post after 6-8 weeks
  Trait and state mindfulness
Alcohol consumption | pre, post after 6-8 weeks, follow-up three months later
  Frequency of drinking days and quantity of alcohol consumed
Dependence Severity (Alcohol Dependence Scale) | pre, post after 6-8 weeks, follow-up three months later
  Craving, urge and dependence severity assessed via questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Beck, Prof. Dr., Principal Investigator — Faculty of Health Sciences, Health and Medical University, University of Potsdam, Potsdam, Germany; Nina Romanczuk-Seiferth, Prof. Dr., Principal Investigator — Department of Psychology, Clinical Psychology and Psychotherapy, MSB Medical School Berlin, Berlin, Germany; Surjo Soekadar, Prof. Dr., Principal Investigator — Department of Psychiatry and Psychotherapy, Charité - Berlin University of Medicine, Berlin, Germany
Locations (1):
- Charité - Berlin University of Medicine, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ekhtiari H, Zare-Bidoky M, Sangchooli A, Janes AC, Kaufman MJ, Oliver JA, Prisciandaro JJ, Wustenberg T, Anton RF, Bach P, Baldacchino A, Beck A, Bjork JM, Brewer J, Childress AR, Claus ED, Courtney KE, Ebrahimi M, Filbey FM, Ghahremani DG, Azbari PG, Goldstein RZ, Goudriaan AE, Grodin EN, Hamilton JP, Hanlon CA, Hassani-Abharian P, Heinz A, Joseph JE, Kiefer F, Zonoozi AK, Kober H, Kuplicki R, Li Q, London ED, McClernon J, Noori HR, Owens MM, Paulus MP, Perini I, Potenza M, Potvin S, Ray L, Schacht JP, Seo D, Sinha R, Smolka MN, Spanagel R, Steele VR, Stein EA, Steins-Loeber S, Tapert SF, Verdejo-Garcia A, Vollstadt-Klein S, Wetherill RR, Wilson SJ, Witkiewitz K, Yuan K, Zhang X, Zilverstand A. A methodological checklist for fMRI drug cue reactivity studies: development and expert consensus. Nat Protoc. 2022 Mar;17(3):567-595. doi: 10.1038/s41596-021-00649-4. Epub 2022 Feb 4. PMID 35121856
- [Background] Swick D, Ashley V, Turken U. Are the neural correlates of stopping and not going identical? Quantitative meta-analysis of two response inhibition tasks. Neuroimage. 2011 Jun 1;56(3):1655-65. doi: 10.1016/j.neuroimage.2011.02.070. Epub 2011 Mar 3. PMID 21376819
- [Background] Kleckner IR, Wormwood JB, Simmons WK, Barrett LF, Quigley KS. Methodological recommendations for a heartbeat detection-based measure of interoceptive sensitivity. Psychophysiology. 2015 Nov;52(11):1432-40. doi: 10.1111/psyp.12503. Epub 2015 Aug 12. PMID 26265009
- [Derived] Rosenthal A, Haslacher D, Garbusow M, Pangratz L, Apfel B, Soekadar S, Romanczuk-Seiferth N, Beck A. Neuromodulation and mindfulness as therapeutic treatment in detoxified patients with alcohol use disorder. BMC Psychiatry. 2024 Sep 27;24(1):635. doi: 10.1186/s12888-024-06085-4. PMID 39334026
- See also: Related Info — http://www.trr265.org/